CLINICAL TRIAL: NCT04394000
Title: Impact of Implementation of an Intensified Thromboprofylaxis Protocol in in Critically Ill ICU Patients With COVID-19: a Longitudinal Controlled Before-after Study
Brief Title: Impact of an Intensified Thromboprofylaxis Protocol in COVID-19
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Jessa_20.48
Record Dates: First submitted 2020-05-16; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: COVID19; Thromboembolism
MeSH Terms: conditions — COVID-19; Thromboembolism | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before or control group: All patients admitted to ICU from March 13th 2020 until March 30th 2020 received routine low dose pharmacological VTE prophylaxis
  Interventions: Other: standard protocol
- After or intervention group: On March 31th 2020 an individualised, more aggressive thromboprophylaxis protocol was implemented. This individualised protocol contains three cornerstones: an increase in dosage of prophylactic LMWH close to therapeutic doses, introduction of routine venous ultrasonography and daily measurements of plasma anti-factor Xa activity
  Interventions: Other: thromboprofylaxis protocol

INTERVENTIONS:
Other: thromboprofylaxis protocol — This individualised protocol contains three cornerstones: an increase in dosage of prophylactic LMWH close to therapeutic doses, introduction of routine venous ultrasonography and daily measurements of plasma anti-factor Xa activity
  Groups: After or intervention group
Other: standard protocol — This protocol contains a routine low dose pharmacological venous thromboembolism (VTE) prophylaxis with LMWH
  Groups: Before or control group

SUMMARY:
The aim of this study is to investigate and compare the mortality, the incidence of DVT and the incidence of kidney and liver failure in patients admitted to the ICU before and after the implementation of an intensified thromboprofylaxis protocol on 31st of March 2020. Patients in the before group are admitted at the ICU from 13/3/2020-30/3/2020 and patients in the after group are admitted to the ICU from 31/3 until 20/4/2020.

DETAILED DESCRIPTION:
Background Patients admitted to the Intensive Care Unit (ICU) are known to be at risk for thrombo-embolic events. Virchow's triad describes the major risk factors in three categories: venous stasis, vessel injury and activation of blood coagulation. A prolonged mechanical ventilation together with the hemodynamic effects of this ventilation with a high positive and expiratory pressure (PEEP), the presence of central venous catheters, the immobilization of these patients and the presence of obesity or other comorbidities can attribute to the occurrence of a deep venous thrombosis (DVT) in patients admitted at ICU. The incidence of DVT during ICU stay has been reported between 5 and 15%.

On the 13th of March, the first COVID-19 patient was admitted at the ICU at the Jessa Hospital. Within a few days, the admissions at our COVID-19 unit grew exponential. In these difficult time, research concerning COVID-19 has been performed indicating the COVID-19 virus induces a hyper-inflammatory state. It has been suggested that systemic inflammation induces endothelial injury. This will activate the coagulation cascade and impair fibrinolysis with disruption of endothelial barrier, and loss of physiologic antithrombotic factors which may elevated the risk for DVTs significantly. Up to now, there is still no causal treatment for COVID-19. The current management of COVID-19 is mainly supportive i.e. a prolonged inflammatory status and a prolonged risk for VTE.

We have shown in a previous cross sectional study that the prevalence of deep venous thrombosis (DVT) in critically ill ICU patients with COVID-19 treated with a prophylactic dose of low molecular weight heparin (LMWH) is more than 60% (submitted manuscript). Consequently, the risk of VTE complications in this patient group is very high. In the light of these findings, an intensified thromboprofylaxis protocol was applied in critically ill ICU patients with COVID-19 at our ICU units since 31st of March 2020.

Aim The aim of this study is to investigate and compare the mortality, the incidence of DVT and the incidence of kidney and liver failure in patients admitted to the ICU before and after the implementation of an intensified thromboprofylaxis protocol on 31st of March 2020. Patients in the before group are admitted at the ICU from 13/3/2020-30/3/2020 and patients in the after group are admitted to the ICU from 31/3 until 20/4/2020.

Design This is a retrospective, longitudinal, before-after controlled study investigating the mortality, the incidence of DVT and the incidence of kidney and liver failure in COVID-19 patients admitted to the ICU before and after the implementation of an intensified thromboprofylaxis protocol.

Outcome measures The primary endpoint of this retrospective study is to investigate the mortality in critically ill ICU patients before and after the implementation of the intensified thromboprofylaxis protocol in our hospital.

Secondary endpoints are the incidence of DVTs with the number and locations of these thromboses, the incidence of kidney failure and the incidence of liver failure in COVID-19 patients admitted to the ICU before and after the implementation of the thromboprofylaxis protocol.

Additional data collection

Additional collected parameters are listed below and are collected as a standard-of-care in our hospital:

* Demographics: i.e age, gender, BMI, Apache II score (to predict mortality)
* Comorbidities: smoking, obesity, hypertension, diabetes, cardiovascular disease, respiratory disease, malignancies, renal failure (AKI), liver failure, gastrointestinal disease, neurological conditions, mental state, other
* Symptoms at the time of admission to ICU: i.e fever, body temperature, dyspnoea, headache, diarrhea etc…
* Laboratory results of all standard parameters measured
* Treatment: antiviral agents, antibiotics, etc…
* Complications: shock, heart failure, sepsis, stroke, etc…
* Ventilation: method, PEEP, FiO2, P/F ratio ..
* SOFA score (Sequential Organ Failure Assessment)
* Radiological findings: pneumonia, ground-glass opacity..

ELIGIBILITY:
Inclusion Criteria:

- All adult COVID19+ patients admitted to the ICU from 13th of March until 20th of April 2020.

Exclusion Criteria:

- Patients younger than 18 years old.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult COVID19+ patients admitted to the ICU from 13th of March until 20th of April 2020.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
2 week mortality | 2 weeks after admission at ICU
  mortality was assessed in all COVID 19 patients admitted to the ICU

SECONDARY OUTCOMES:
incidence of venous thromboembolism | during ICU stay up till 3th of May 2020
  the incidence of venous thromboembolism was evaluated in all COVID 19 patients admitted to the ICU
1 week mortality | 1 week after admission at ICU
  mortality was assessed in all COVID 19 patients admitted to the ICU
3 week mortality | 3 weeks after admission at ICU
  mortality was assessed in all COVID 19 patients admitted to the ICU
1 month mortality | 1 month after admission at ICU
  mortality was assessed in all COVID 19 patients admitted to the ICU
incidence of kidney failure | during ICU stay up till 3th of May 2020
  incidence of acute kidney failure in all COVID 19 patients admitted to the ICU
incidence of continuous renal replacement therapy (CRRT) | during ICU stay up till 3th of May 2020
  incidence of continuous renal replacement therapy (CRRT) in all COVID 19 patients admitted to the ICU
lowest PaO2/FiO2 (P/F) ratio | during ICU stay up till 3th of May 2020
  evaluation of the lowest P/F ratio in all COVID 19 patients admitted to the ICU
highest Sequential Organ Failure Assessment (SOFA) score | during ICU stay up till 3th of May 2020
  evaluation of the highest SOFA score in all COVID 19 patients admitted to the ICU
length of stay | during ICU and hospital stay up till 3th of May 2020
  evaluation of the length of stay in ICU and hospital of all COVID 19 patients admitted to the ICU
highest bilirubin | during ICU stay up till 3th of May 2020
  evaluation of the highest bilirubine level in all COVID 19 patients admitted to the ICU
highest ( AST | during ICU stay up till 3th of May 2020
  evaluation of the highest AST level in all COVID 19 patients admitted to the ICU
highest Aspartaat-Amino-Transferase (ALT) | during ICU stay up till 3th of May 2020
  evaluation of the highest ALT level in all COVID 19 patients admitted to the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stessel B, Vanvuchelen C, Bruckers L, Geebelen L, Callebaut I, Vandenbrande J, Pellens B, Van Tornout M, Ory JP, van Halem K, Messiaen P, Herbots L, Ramaekers D, Dubois J. Impact of implementation of an individualised thromboprophylaxis protocol in critically ill ICU patients with COVID-19: A longitudinal controlled before-after study. Thromb Res. 2020 Oct;194:209-215. doi: 10.1016/j.thromres.2020.07.038. Epub 2020 Jul 22. PMID 32788120